CLINICAL TRIAL: NCT06450405
Title: Androgen Effects on the Reproductive Neuroendocrine Axis
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: The study sponsor terminated the grant funding.
Sponsor: University of California, San Diego (Other)
Collaborators: National Institutes of Health (NIH) (NIH); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Antoni Duleba, Professor, University of California, San Diego
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 808679; 1R01HD111650-01 (NIH)
Record Dates: First submitted 2024-04-30; First posted 2024-06-10 (Actual); Results first posted 2025-07-14 (Actual); Last update posted 2025-07-22 (Actual); Status verified 2025-07

CONDITIONS: Transgenderism; Reproductive Issues
MeSH Terms: conditions — Transsexualism | interventions — testosterone 17 beta-cypionate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- TGM initiating TRT (Active Comparator): Transgender men/non-binary/non-gender-conforming initiating testosterone replacement therapy
  Interventions: Drug: Testosterone Cypionate 50 MG/ML Injectable Solution
- CGF control group (No Intervention): Cisgender females serving as a control group

INTERVENTIONS:
Drug: Testosterone Cypionate 50 MG/ML Injectable Solution — Participants in the initiating group will receive weekly doses of testosterone for gender-affirming care.
  Other Names: Testosterone Replacement Therapy
  Arms: TGM initiating TRT

SUMMARY:
This research study investigates whether male-level exogenous androgens inhibit the reproductive neuroendocrine axis in otherwise healthy (non-PCOS) females.

DETAILED DESCRIPTION:
Testosterone Replacement Therapy (TRT) is the mainstay of gender affirming care for transgender men (TGM) who have male gender identity after female sex assignment at birth. TGM receiving TRT over time exhibit irregular menstrual bleeding, however, the mechanism of menstrual disruption is unknown. Therefore, the investigators propose to evaluate the effect of chronic testosterone (T) exposure on ovarian hormones and pituitary gonadotropin release that determines menstrual cyclicity. The investigators will conduct a detailed study of blood reproductive hormone secretion in TGM before and during TRT as well as in untreated cisgender female (CGF) control subjects who report female gender identity congruent with female sex assignment at birth. The investigators will also perform periodic clinical and ultrasonographic evaluations.

ELIGIBILITY:
Inclusion Criteria: Transgender/Non-binary Group, Initiating Testosterone Group

* Provision of signed and dated informed consent form
* Stated willingness to comply with all study procedures and availability for the duration of the study
* Aged 18-35
* Plan to initiate testosterone therapy
* History of regular menstrual cycles (every 24-35 days) at baseline, before beginning TRT

Inclusion Criteria: Cisgender Female Group

* Provision of signed and dated informed consent form
* Stated willingness to comply with all study procedures and availability for the duration of the study
* Aged 18-35
* Having regular menstrual cycles (every 24-35 days)

Exclusion Criteria: All

* Pregnant
* Incarcerated
* Known cognitive impairment or institutionalized
* Hemoglobin less than 11 gm/dl at screening evaluation
* Weight less than 110 pounds
* BMI <18 or >35
* Current endocrine disease- including untreated thyroid abnormalities, pituitary or adrenal disease, polycystic ovary syndrome, or androgen producing tumor
* Current or recent pregnancy within two months of study enrollment
* Current or recent breast feeding within two months of study enrollment
* Diabetes, or renal, liver, or heart disease
* History of oophorectomy or hysterectomy
* History of radiation or surgery involving brain structures and/or pelvis/pelvic organs
* Currently taking any medications that may affect their reproductive hormones, such as contraceptive medications, androgens, estrogens, progestins, GnRH antagonists, GnRH agonists, insulinomimetics, and metformin.
* History of prior testosterone therapy

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Cisgender females; Transgender males/non-binary/gender non-conforming initiating testosterone replacement therapy
Enrollment: 2 (Actual)
Dates: Start 2025-02-26 (Actual); Primary Completion 2025-02-26 (Actual); Study Completion 2025-03-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Antoni Duleba, MD, Principal Investigator — UC San Diego
Locations (1):
- University of California San Diego, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: No
We will not be sharing IPD.

REFERENCES:
- [Background] Coleman E, Radix AE, Bouman WP, Brown GR, de Vries ALC, Deutsch MB, Ettner R, Fraser L, Goodman M, Green J, Hancock AB, Johnson TW, Karasic DH, Knudson GA, Leibowitz SF, Meyer-Bahlburg HFL, Monstrey SJ, Motmans J, Nahata L, Nieder TO, Reisner SL, Richards C, Schechter LS, Tangpricha V, Tishelman AC, Van Trotsenburg MAA, Winter S, Ducheny K, Adams NJ, Adrian TM, Allen LR, Azul D, Bagga H, Basar K, Bathory DS, Belinky JJ, Berg DR, Berli JU, Bluebond-Langner RO, Bouman MB, Bowers ML, Brassard PJ, Byrne J, Capitan L, Cargill CJ, Carswell JM, Chang SC, Chelvakumar G, Corneil T, Dalke KB, De Cuypere G, de Vries E, Den Heijer M, Devor AH, Dhejne C, D'Marco A, Edmiston EK, Edwards-Leeper L, Ehrbar R, Ehrensaft D, Eisfeld J, Elaut E, Erickson-Schroth L, Feldman JL, Fisher AD, Garcia MM, Gijs L, Green SE, Hall BP, Hardy TLD, Irwig MS, Jacobs LA, Janssen AC, Johnson K, Klink DT, Kreukels BPC, Kuper LE, Kvach EJ, Malouf MA, Massey R, Mazur T, McLachlan C, Morrison SD, Mosser SW, Neira PM, Nygren U, Oates JM, Obedin-Maliver J, Pagkalos G, Patton J, Phanuphak N, Rachlin K, Reed T, Rider GN, Ristori J, Robbins-Cherry S, Roberts SA, Rodriguez-Wallberg KA, Rosenthal SM, Sabir K, Safer JD, Scheim AI, Seal LJ, Sehoole TJ, Spencer K, St Amand C, Steensma TD, Strang JF, Taylor GB, Tilleman K, T'Sjoen GG, Vala LN, Van Mello NM, Veale JF, Vencill JA, Vincent B, Wesp LM, West MA, Arcelus J. Standards of Care for the Health of Transgender and Gender Diverse People, Version 8. Int J Transgend Health. 2022 Sep 6;23(Suppl 1):S1-S259. doi: 10.1080/26895269.2022.2100644. eCollection 2022. PMID 36238954
- [Background] Hembree WC, Cohen-Kettenis PT, Gooren L, Hannema SE, Meyer WJ, Murad MH, Rosenthal SM, Safer JD, Tangpricha V, T'Sjoen GG. Endocrine Treatment of Gender-Dysphoric/Gender-Incongruent Persons: An Endocrine Society Clinical Practice Guideline. J Clin Endocrinol Metab. 2017 Nov 1;102(11):3869-3903. doi: 10.1210/jc.2017-01658. PMID 28945902
- [Background] Deutsch MB, Bhakri V, Kubicek K. Effects of cross-sex hormone treatment on transgender women and men. Obstet Gynecol. 2015 Mar;125(3):605-610. doi: 10.1097/AOG.0000000000000692. PMID 25730222
- [Background] McFarland J, Craig W, Clarke NJ, Spratt DI. Serum Testosterone Concentrations Remain Stable Between Injections in Patients Receiving Subcutaneous Testosterone. J Endocr Soc. 2017 Jul 21;1(8):1095-1103. doi: 10.1210/js.2017-00148. eCollection 2017 Aug 1. PMID 29264562
- [Background] Nakamura A, Watanabe M, Sugimoto M, Sako T, Mahmood S, Kaku H, Nasu Y, Ishii K, Nagai A, Kumon H. Dose-response analysis of testosterone replacement therapy in patients with female to male gender identity disorder. Endocr J. 2013;60(3):275-81. doi: 10.1507/endocrj.ej12-0319. Epub 2012 Oct 27. PMID 23117148
- [Background] Conron KJ, Scott G, Stowell GS, Landers SJ. Transgender health in Massachusetts: results from a household probability sample of adults. Am J Public Health. 2012 Jan;102(1):118-22. doi: 10.2105/AJPH.2011.300315. Epub 2011 Nov 28. PMID 22095354
- [Background] Clark TC, Lucassen MF, Bullen P, Denny SJ, Fleming TM, Robinson EM, Rossen FV. The health and well-being of transgender high school students: results from the New Zealand adolescent health survey (Youth'12). J Adolesc Health. 2014 Jul;55(1):93-9. doi: 10.1016/j.jadohealth.2013.11.008. Epub 2014 Jan 14. PMID 24438852
- [Background] Kuyper L, Wijsen C. Gender identities and gender dysphoria in the Netherlands. Arch Sex Behav. 2014 Feb;43(2):377-85. doi: 10.1007/s10508-013-0140-y. Epub 2013 Jul 16. PMID 23857516
- [Background] Van Caenegem E, Wierckx K, Elaut E, Buysse A, Dewaele A, Van Nieuwerburgh F, De Cuypere G, T'Sjoen G. Prevalence of Gender Nonconformity in Flanders, Belgium. Arch Sex Behav. 2015 Jul;44(5):1281-7. doi: 10.1007/s10508-014-0452-6. Epub 2015 Jan 15. PMID 25588709
- [Background] Meerwijk EL, Sevelius JM. Transgender Population Size in the United States: a Meta-Regression of Population-Based Probability Samples. Am J Public Health. 2017 Feb;107(2):e1-e8. doi: 10.2105/AJPH.2016.303578. PMID 28075632
- [Background] Meyer IH, Brown TN, Herman JL, Reisner SL, Bockting WO. Demographic Characteristics and Health Status of Transgender Adults in Select US Regions: Behavioral Risk Factor Surveillance System, 2014. Am J Public Health. 2017 Apr;107(4):582-589. doi: 10.2105/AJPH.2016.303648. Epub 2017 Feb 16. PMID 28207334
- [Background] De Cuypere G, Van Hemelrijck M, Michel A, Carael B, Heylens G, Rubens R, Hoebeke P, Monstrey S. Prevalence and demography of transsexualism in Belgium. Eur Psychiatry. 2007 Apr;22(3):137-41. doi: 10.1016/j.eurpsy.2006.10.002. Epub 2006 Dec 26. PMID 17188846
- [Background] Zucker KJ, Lawrence AA. Epidemiology of Gender Identity Disorder: Recommendations for the Standards of Care of the World Professional Association for Transgender Health. Int J Transgenderism. 2009;11(1):8-18. doi:10.1080/15532730902799946
- [Background] Coleman E, Bockting W, Botzer M, et al. Standards of Care for the Health of Transsexual, Transgender, and Gender-Nonconforming People, Version 7. Int J Transgenderism. 2012;13(4):165-232. doi:10.1080/15532739.2011.700873
- [Background] Spinder T, Spijkstra JJ, van den Tweel JG, Burger CW, van Kessel H, Hompes PG, Gooren LJ. The effects of long term testosterone administration on pulsatile luteinizing hormone secretion and on ovarian histology in eugonadal female to male transsexual subjects. J Clin Endocrinol Metab. 1989 Jul;69(1):151-7. doi: 10.1210/jcem-69-1-151. PMID 2471710
- [Background] Pelusi C, Costantino A, Martelli V, Lambertini M, Bazzocchi A, Ponti F, Battista G, Venturoli S, Meriggiola MC. Effects of three different testosterone formulations in female-to-male transsexual persons. J Sex Med. 2014 Dec;11(12):3002-11. doi: 10.1111/jsm.12698. Epub 2014 Sep 24. PMID 25250780
- [Background] Mueller A, Kiesewetter F, Binder H, Beckmann MW, Dittrich R. Long-term administration of testosterone undecanoate every 3 months for testosterone supplementation in female-to-male transsexuals. J Clin Endocrinol Metab. 2007 Sep;92(9):3470-5. doi: 10.1210/jc.2007-0746. Epub 2007 Jun 19. PMID 17579193
- [Background] Moravek MB, Kinnear HM, George J, Batchelor J, Shikanov A, Padmanabhan V, Randolph JF. Impact of Exogenous Testosterone on Reproduction in Transgender Men. Endocrinology. 2020 Mar 1;161(3):bqaa014. doi: 10.1210/endocr/bqaa014. PMID 32105330
- [Background] Wierckx K, Van Caenegem E, Pennings G, Elaut E, Dedecker D, Van de Peer F, Weyers S, De Sutter P, T'Sjoen G. Reproductive wish in transsexual men. Hum Reprod. 2012 Feb;27(2):483-7. doi: 10.1093/humrep/der406. Epub 2011 Nov 28. PMID 22128292
- [Background] Cipres D, Seidman D, Cloniger C 3rd, Nova C, O'Shea A, Obedin-Maliver J. Contraceptive use and pregnancy intentions among transgender men presenting to a clinic for sex workers and their families in San Francisco. Contraception. 2017 Feb;95(2):186-189. doi: 10.1016/j.contraception.2016.09.005. Epub 2016 Sep 9. PMID 27621044
- [Background] Moseson H, Fix L, Hastings J, Stoeffler A, Lunn MR, Flentje A, Lubensky ME, Capriotti MR, Ragosta S, Forsberg H, Obedin-Maliver J. Pregnancy intentions and outcomes among transgender, nonbinary, and gender-expansive people assigned female or intersex at birth in the United States: Results from a national, quantitative survey. Int J Transgend Health. 2021 Nov 17;22(1-2):30-41. doi: 10.1080/26895269.2020.1841058. eCollection 2021. PMID 34796363
- [Background] Kerman HM, Pham A, Crouch JM, Albertson K, Salehi P, Inwards-Breland DJ, Ahrens KR. Gender Diverse Youth on Fertility and Future Family: A Qualitative Analysis. J Adolesc Health. 2021 Jun;68(6):1112-1120. doi: 10.1016/j.jadohealth.2021.01.002. Epub 2021 Mar 10. PMID 33712381
- [Background] Rafferty J; COMMITTEE ON PSYCHOSOCIAL ASPECTS OF CHILD AND FAMILY HEALTH; COMMITTEE ON ADOLESCENCE; SECTION ON LESBIAN, GAY, BISEXUAL, AND TRANSGENDER HEALTH AND WELLNESS. Ensuring Comprehensive Care and Support for Transgender and Gender-Diverse Children and Adolescents. Pediatrics. 2018 Oct;142(4):e20182162. doi: 10.1542/peds.2018-2162. Epub 2018 Sep 17. PMID 30224363
- [Background] Light A, Wang LF, Zeymo A, Gomez-Lobo V. Family planning and contraception use in transgender men. Contraception. 2018 Oct;98(4):266-269. doi: 10.1016/j.contraception.2018.06.006. Epub 2018 Jun 23. PMID 29944875
- [Background] Light AD, Obedin-Maliver J, Sevelius JM, Kerns JL. Transgender men who experienced pregnancy after female-to-male gender transitioning. Obstet Gynecol. 2014 Dec;124(6):1120-1127. doi: 10.1097/AOG.0000000000000540. PMID 25415163
- [Background] Taub RL, Ellis SA, Neal-Perry G, Magaret AS, Prager SW, Micks EA. The effect of testosterone on ovulatory function in transmasculine individuals. Am J Obstet Gynecol. 2020 Aug;223(2):229.e1-229.e8. doi: 10.1016/j.ajog.2020.01.059. Epub 2020 Feb 8. PMID 32044312
- [Background] Dewis P, Newman M, Ratcliffe WA, Anderson DC. Does testosterone affect the normal menstrual cycle? Clin Endocrinol (Oxf). 1986 May;24(5):515-21. doi: 10.1111/j.1365-2265.1986.tb03280.x. PMID 3098455
- [Background] Scheele F, Hompes PG, Gooren LJ, Spijkstra JJ, Spinder T. The effect of 6 weeks of testosterone treatment on pulsatile luteinizing hormone secretion in eugonadal female-to-male transsexuals. Fertil Steril. 1991 Mar;55(3):608-11. doi: 10.1016/s0015-0282(16)54194-6. PMID 2001760
- [Background] Ropelato MG, Rudaz MC, Escobar ME, Bengolea SV, Calcagno ML, Veldhuis JD, Barontini M. Acute effects of testosterone infusion on the serum luteinizing hormone profile in eumenorrheic and polycystic ovary syndrome adolescents. J Clin Endocrinol Metab. 2009 Sep;94(9):3602-10. doi: 10.1210/jc.2009-0402. Epub 2009 Jun 30. PMID 19567528
- [Background] Spinder T, Spijkstra JJ, Gooren LJ, Hompes PG, van Kessel H. Effects of long-term testosterone administration on gonadotropin secretion in agonadal female to male transsexuals compared with hypogonadal and normal women. J Clin Endocrinol Metab. 1989 Jan;68(1):200-7. doi: 10.1210/jcem-68-1-200. PMID 2491861
- [Background] T'Sjoen G, Arcelus J, Gooren L, Klink DT, Tangpricha V. Endocrinology of Transgender Medicine. Endocr Rev. 2019 Feb 1;40(1):97-117. doi: 10.1210/er.2018-00011. PMID 30307546
- [Background] Mwamba RN, Ekwonu A, Guimaraes PVB, Raheem OA. The efficacy, safety, and outcomes of testosterone use among transgender men patients: A review of the literature. Neurourol Urodyn. 2023 Jun;42(5):921-930. doi: 10.1002/nau.25094. Epub 2022 Nov 20. PMID 36403286
- [Background] Kassam A, Overstreet JW, Snow-Harter C, De Souza MJ, Gold EB, Lasley BL. Identification of anovulation and transient luteal function using a urinary pregnanediol-3-glucuronide ratio algorithm. Environ Health Perspect. 1996 Apr;104(4):408-13. doi: 10.1289/ehp.96104408. PMID 8732951
- [Background] Santoro N, Crawford SL, Allsworth JE, Gold EB, Greendale GA, Korenman S, Lasley BL, McConnell D, McGaffigan P, Midgely R, Schocken M, Sowers M, Weiss G. Assessing menstrual cycles with urinary hormone assays. Am J Physiol Endocrinol Metab. 2003 Mar;284(3):E521-30. doi: 10.1152/ajpendo.00381.2002. Epub 2002 Nov 19. PMID 12441312
- [Background] Pfizer Inc. Depo®-Testosterone (testosterone cypionate injection, USP0 [package insert]. U.S. Food and Drug Administration website. https://www.accessdata.fda.gov/drugsatfda_docs/label/2014/085635s029lbl.pdf. Accessed May 30, 2022.
- See also: Pfizer Inc. Depo®-Testosterone (testosterone cypionate injection, USP0 [package insert]. U.S. Food and Drug Administration website. — https://www.accessdata.fda.gov/drugsatfda_docs/label/2014/085635s029lbl.pdf

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The researchers enrolled 2 cisgender female participants before the study was terminated. Enrolled CGFs signed consent forms, but did not participate in any study activities. There is no analyzable data.
Period: Overall Study
Arm/Group | TGM Initiating TRT | CGF Control Group
Started | 0 | 2
Completed | 0 | 0
Not Completed | 0 | 2
Not completed — Study funding terminated. | 0 | 2

BASELINE CHARACTERISTICS:
Population: The study terminated before enrollment of TGM initiating TRT. Two CGF participants signed the consent form, but did not provide any demographic information. The only data we collected were name and signature. No data were analyzed. No data will be analyzed in the future. The enrollees would have been scheduled for study visits a week or two after signing the consent form.
Groups:
- Total: Total of all reporting groups
Arm/Group | TGM Initiating TRT | CGF Control Group | Total
Number analyzed (Participants) | 0 | 0 | 0
Age, Categorical
Age, Continuous [unit: years]
Sex: Female, Male
Race (NIH/OMB)
Region of Enrollment

OUTCOME MEASURES:

1. Primary Outcome: Evidence of Luteal Activity (ELA)
Description: Evidence of Luteal Activity (ELA), as defined by serum progesterone level above 3 ng/mL in transgender men initiating testosterone replacement therapy.
Time Frame: Through study completion, an average of 7 months.
Population: The study sponsor terminated the grant funding before any data, besides names and signatures on consent forms, were collected. There are no data to analyze. No data will be analyzed in the future.
Arm/Group | TGM Initiating TRT | CGF Control Group
Number analyzed (Participants) | 0 | 0

2. Primary Outcome: Determination of Pulsatile LH Secretion
Description: Subjects will have baseline measurement of serum LH immediately followed by frequent blood sampling at 10-min intervals for 8 h. We will measure LH pulse frequency, the number of LH pulses per 8 hours.
Time Frame: Through study completion, an average of 7 months.
Population: as for outcome 1
Arm/Group | TGM Initiating TRT | CGF Control Group
Number analyzed (Participants) | 0 | 0

3. Primary Outcome: Uterine Bleeding Pattern.
Description: All subjects will complete a daily uterine bleeding log using REDCap®
Time Frame: Through study completion, an average of 7 months.
Population: as for outcome 1
Arm/Group | TGM Initiating TRT | CGF Control Group
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Evaluate Serum Reproductive Hormones
Description: Measurement of serum FSH, AMH, LH, estradiol, and testosterone levels
Time Frame: Through study completion, an average of 7 months.
Population: as for outcome 1
Arm/Group | TGM Initiating TRT | CGF Control Group
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: There is no time frame because the study sponsor terminated the grant funding before any analyzable data were collected. The study sponsor terminated the grant funding days after the first two participants signed consent forms, but before any data, besides names and signatures on consent forms, were collected. There are no data to analyze. No data will be analyzed in the future.
Description: There was no adverse event collection timeframe because the two enrollees did not have any study visits. The study sponsor terminated the grant funding before any data, besides names and signatures on consent forms, were collected. There are no adverse event data to collect or to analyze.
Arm/Group | TGM Initiating TRT | CGF Control Group
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-09-04): https://cdn.clinicaltrials.gov/large-docs/05/NCT06450405/Prot_SAP_000.pdf